CLINICAL TRIAL: NCT05848245
Title: Reducing Aerosol And Bioaerosol Using Different Oral Suctions In Dental Clinic, Randomized Clinical Trial
Brief Title: Reducing Aerosol and Bioaerosol Using Different Oral Suctions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Zuhair Saleh Natto, Associate professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 351-12-21
Record Dates: First submitted 2023-04-14; First posted 2023-05-08 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Infections; Oral Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- low suction (Experimental): It is a small and narrow in diameter help to remove saliva , blood and debris and provide a clear vision to healthcare worker. It will be used as conventional way; low suction will be hanged on patient mouth and moved it thoroughly as needed it, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Interventions: Device: low suction
- intraoral suction (Active Comparator): Intraoral suction is attached to high volume excavation hose and provide continuous suction with a bite block, tongue, and oral pathway protection.It will be used as conventional way; intraoral suction will be hanged on patient mouth and moved it thoroughly as needed it, high suction will be moved with scaler, and extraoral suction where on right hand side of patient, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Interventions: Device: intraoral suction
- high & low suction (Experimental): Low section is a small and narrow in diameter help to remove saliva , blood and debris and provide a clear vision to healthcare worker.
  High section is a large tube designed to suction large amount of air volume and droplet. It will be used as conventional way; low suction will be hanged on patient mouth and moved it thoroughly as needed it, high suction will be moved with scaler, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Interventions: Device: high & low suction
- extra-oral suction & low suction (Experimental): EOS is used to remove aerosol and droplet that arising from patient mouth and filtering air. The device starts from air volume level 1 to level 10.
  Low section is a small and narrow in diameter help to remove saliva , blood and debris and provide a clear vision to healthcare worker. It will be used as conventional way; low suction will be hanged on patient mouth and moved it thoroughly as needed it, and extraoral suction where on right hand side of patient, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Interventions: Device: extra-oral suction & low suction
- extra-oral suction and intraoral suction (Experimental): EOS is used to remove aerosol and droplet that arising from patient mouth and filtering air. The device starts from air volume level 1 to level 10.
  High section is a large tube designed to suction large amount of air volume and droplet. It will be used as conventional way; intraoral suction will be hanged on patient mouth and moved it thoroughly as needed it, and extraoral suction where on right hand side of patient, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Interventions: Device: Extra-Oral Suction and Intraoral Suction

INTERVENTIONS:
Device: low suction — This group receives low-volume intraoral suction during procedures. Low suction typically refers to standard saliva ejectors, which provide minimal suction power and are commonly used in routine dental treatments.
  Arms: low suction
Device: intraoral suction — This group receives conventional intraoral suction, likely using high-volume evacuators (HVE), which are more effective than low suction. This arm serves as the comparison or standard-of-care group against which other interventions are evaluated.
  Arms: intraoral suction
Device: high & low suction — Participants in this group receive both high-volume and low-volume intraoral suction simultaneously. The combined use aims to optimize fluid and aerosol control, with high suction capturing larger volumes and low suction assisting in continuous evacuation.
  Arms: high & low suction
Device: extra-oral suction & low suction — This group receives a combination of extra-oral suction (a device placed outside the mouth to capture aerosols at the source) and low-volume intraoral suction. This setup is designed to reduce airborne particles during procedures by controlling both intraoral and environmental aerosols.
  Arms: extra-oral suction & low suction
Device: Extra-Oral Suction and Intraoral Suction — This group is treated using both extra-oral suction and intraoral suction, likely high-volume. The dual approach targets aerosol containment both at the oral cavity level and in the surrounding air, representing a comprehensive strategy for infection control during aerosol-generating procedures.
  Arms: extra-oral suction and intraoral suction

SUMMARY:
Aerosol particles generated when using dental instrument such as ultrasonic and high air driven handpieces, this aerosol is mixture of blood, saliva, infectious agents, and dental materials. Inhaler dust that range between PM2.5 to PM10 could transferred to the human lung's terminal bronchioles and alveoli that cause a harm effect. The aim of this study to assess the effectiveness of different dental suction devices that could be contributed to decrease risk of particles count, Bacterial and fungal that arising from patient mouth to indoor air dental clinic. This is a randomized clinical trial will be conducted in three different places: educational hospital, public hospital, and private clinic. In each place 40 subject will be recruited. Measurement including particles count and microorganism will be taken before 15 minutes and during of scaling and prophylaxis procedure to measure particles count, oral bacteria, fungus, and microbial air. In this study will be compared between four intervention groups; Group A with high and low suction only, Group B using dry shield suction and low section, Group C using extra-oral suction with high and low suction, and Group D using dry shield suction and extra-oral suction and low section. Difference between each categorical groups and particle, oral bacterial, fungus, and microbial air concentration will be tested using two-way ANOVA test or one way ANOVA test. Statistical analysis will be carried using STATA version 13.

DETAILED DESCRIPTION:
Aerosols described as any fluid and solid particles dropped in the air. Any particles less than 50 micrometer in diameter could be suspended into air for extended period before rest on environmental surfaces or enter respiratory tract. Bioaerosol are a complex mixture of airborne particles of biological origin such as bacteria, viruses, and fungus.

In dental clinic, dental team are exposed to infectious droplet through a direct contact with body fluid of patient, contact with environmental surfaces or instrument. Dental aerosol might be not easily to measure. However, many studies assess the amount of bacteria using bacteria growth media such as blood agar culture. In addition, particle number concentrations are considered as indication for health exposure risk to describe cleanroom. Particles in the range of 0.5-10 µm diameter can be inhaled and held on the human lung's terminal bronchioles and alveoli. Dental instruments and procedure generate varies air-borne contamination amount, the highest bacterial growth was produced by ultra-sonic scaler, followed by the air-driven high-speed handpiece, the air polisher and various other instruments such as the airwater syringe and prophylaxis angles. In addition, one of study in vitro was found the high amount of aerosol and spatter generated from ultrasonic scalar if used without cooling and presence of small amounts of liquid placed at the operative site to mimic blood and saliva.

Using personal protective barrier (PPE) would be prevented spatter droplets but particles which is less than 50 micrometer that consist of infectious agent has the potential to enter the respiratory tract through leaks in masks. The exact hazard effects of dental aerosol not possible to recognize currently however the probable spread of infection should be minimized and eliminated.

Infection control should be carried out to maximum level to provide safe environment in dental clinic. Controlling of aerosol and bioaerosol that generated through a different procedure is important to patient and dental staff in order to reduce transmission of infectious disease through direct contact with a surface prior to aerosol and bioaerosol settle down or through inhalation route.

ELIGIBILITY:
Inclusion criteria

* Adult healthy patient above 18 years of age
* Has scheduled an appointment at dental hygienist clinic for scaling procedure.
* Has at least one score 2 or 3 in one sextant according to community periodontal index of treatment needs (CPITN).

Exclusion criteria

* Number of teeth less than 20 teeth
* Presence of soft or hard tissue lesions
* Pregnant women
* Orthodontic patient
* Partial denture wearer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zuhair Natto, Principal Investigator — King Abdulaziz University
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any IPD with other researchers

REFERENCES:
- [Derived] Bannan A, Kamal I, Al Makishah NH, Natto ZS. Reducing microbial airborne contamination and particulate matter using different oral suctions in dental clinic: A randomized controlled clinical trial. Saudi Dent J. 2024 Feb;36(2):374-380. doi: 10.1016/j.sdentj.2023.11.029. Epub 2023 Nov 28. PMID 38419981

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Suction | Intraoral Suction | High & Low Suction | Extra-oral Suction & Low Suction | Extra-oral Suction and Intraoral Suction
Started | 10 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Suction | Intraoral Suction | High & Low Suction | Extra-oral Suction & Low Suction | Extra-oral Suction and Intraoral Suction | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.4 (6.7) | 32.8 (5.4) | 31 (10.8) | 36.9 (7.6) | 31.4 (9) | 34.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 4 | 3 | 8 | 21
  Male | 9 | 5 | 6 | 7 | 2 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
microbial airborne contamination level [Mean (Standard Deviation); unit: CFU m -3] | 28.4 (14.1) | 28.7 (15.0) | 56.3 (39.2) | 56.8 (35.6) | 31.2 (10.8) | 42.6 (28.3)
Particulate matter [Mean (Standard Deviation); unit: micrograms per cubic meter (µg/m³)] | 121.3 (12.6) | 135.1 (33.8) | 147.6 (30.2) | 128.4 (22.3) | 136.9 (29.9) | 133.9 (27.2)

OUTCOME MEASURES:

1. Primary Outcome: Particulate Matter (PM)
Description: Amount of particulate matter will be measured using Digital dust monitor (model 3443, KANOMAX.USA INC., made in Japan). This device measure particle size that ranges from 0.1 to 10 µm using light scattering method (semiconductor laser radiation light source ) with flow rate of 1 L/min. air is collect through a filter which is built-in in order to eliminate coarse partials.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: micrograms per cubic meter (µg/m³)
Arm/Group | Low Suction | Intraoral Suction | High & Low Suction | Extra-oral Suction & Low Suction | Extra-oral Suction and Intraoral Suction
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
micrograms per cubic meter (µg/m³) | 121.3 (12.6) | 135.1 (33.8) | 147.6 (30.2) | 128.4 (22.3) | 136.9 (29.9)

2. Primary Outcome: Microbial Count
Description: Amount of microbial contamination level. Active air sampler method will be used to collect microorganism onto solid media with flow rate 100 L/ min and lower d50 is 0.5µm. It contains 258 holes with diameter 0.7 mm. Positive hole correction should be used in order to adjust number of colonies forming units per volume of air (CFU m-3) according to the manual.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: CFU/m³
Arm/Group | Low Suction | Intraoral Suction | High & Low Suction | Extra-oral Suction & Low Suction | Extra-oral Suction and Intraoral Suction
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
CFU/m³ | 1117 (624.1) | 325.1 (336.2) | 100.2 (88.3) | 74.2 (28.3) | 45.6 (14.7)

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Low Suction: It is a small and narrow in diameter help to remove saliva , blood and debris and provide a clear vision to healthcare worker. It will be used as conventional way; low suction will be hanged on patient mouth and moved it thoroughly as needed it, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Suction: Dental sections are used to absorb aerosol particles generated when using dental instrument such as ultrasonic and high air driven handpieces, this aerosol is mixture of blood, saliva, infectious agents, and dental materials.
- Intraoral Suction: Intraoral suction is attached to high volume excavation hose and provide continuous suction with a bite block, tongue, and oral pathway protection.It will be used as conventional way; intraoral suction will be hanged on patient mouth and moved it thoroughly as needed it, high suction will be moved with scaler, and extraoral suction where on right hand side of patient, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Suction: Dental sections are used to absorb aerosol particles generated when using dental instrument such as ultrasonic and high air driven handpieces, this aerosol is mixture of blood, saliva, infectious agents, and dental materials.
- High & Low Suction: Low section is a small and narrow in diameter help to remove saliva , blood and debris and provide a clear vision to healthcare worker.
  High section is a large tube designed to suction large amount of air volume and droplet. It will be used as conventional way; low suction will be hanged on patient mouth and moved it thoroughly as needed it, high suction will be moved with scaler, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Suction: Dental sections are used to absorb aerosol particles generated when using dental instrument such as ultrasonic and high air driven handpieces, this aerosol is mixture of blood, saliva, infectious agents, and dental materials.
- Extra-oral Suction & Low Suction: EOS is used to remove aerosol and droplet that arising from patient mouth and filtering air. The device starts from air volume level 1 to level 10.
  Low section is a small and narrow in diameter help to remove saliva , blood and debris and provide a clear vision to healthcare worker. It will be used as conventional way; low suction will be hanged on patient mouth and moved it thoroughly as needed it, and extraoral suction where on right hand side of patient, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Suction: Dental sections are used to absorb aerosol particles generated when using dental instrument such as ultrasonic and high air driven handpieces, this aerosol is mixture of blood, saliva, infectious agents, and dental materials.
- Extra-oral Suction and Intraoral Suction: EOS is used to remove aerosol and droplet that arising from patient mouth and filtering air. The device starts from air volume level 1 to level 10.
  High section is a large tube designed to suction large amount of air volume and droplet. It will be used as conventional way; intraoral suction will be hanged on patient mouth and moved it thoroughly as needed it, and extraoral suction where on right hand side of patient, power will be turned on to level 10, and suction cone will be facing patient mouth and it was away from its around 10 -15 cm based on the manufacturer instruction and to allow comfortable movement of the dental hygienist's hand.
  Suction: Dental sections are used to absorb aerosol particles generated when using dental instrument such as ultrasonic and high air driven handpieces, this aerosol is mixture of blood, saliva, infectious agents, and dental materials.
Arm/Group | Low Suction | Intraoral Suction | High & Low Suction | Extra-oral Suction & Low Suction | Extra-oral Suction and Intraoral Suction
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT05848245/Prot_SAP_000.pdf